CLINICAL TRIAL: NCT06594705
Title: Transcatheter Aortic Valve Replacement Using the JenaValve TrilogyTM Heart Valve System for Clinically Significant Aortic Regurgitation in Patients With Left Ventricular Assist Devices (LVAD)
Brief Title: The JenaValve ALIGN-AR LVAD Registry
Acronym: JENA-VAD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: JenaValve Technology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JVT24002
Record Dates: First submitted 2024-08-29; First posted 2024-09-19 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-07

CONDITIONS: Aortic Regurgitation; Aortic Valve Insufficiency; Aortic Insufficiency; Aortic Valve Disease; Left Ventricular Dysfunction
MeSH Terms: conditions — Aortic Valve Insufficiency; Aortic Valve Disease; Ventricular Dysfunction, Left

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- TAVR in LVAD Patients (Experimental): Transcatheter Aortic Valve Replacement (TAVR)
  TAVR in patients with continuous flow left ventricular assist devices (cfLVAD) and clinically significant aortic regurgitation (AR)
  Interventions: Device: JenaValve Trilogy Heart Valve System

INTERVENTIONS:
Device: JenaValve Trilogy Heart Valve System — TAVR with JenaValve Trilogy Heart Valve System

SUMMARY:
To evaluate the safety and effectiveness of the JenaValve Trilogy™ Heart Valve System for transcatheter aortic valve replacement (TAVR) in subjects with continuous flow left ventricular assist devices (cfLVAD) and clinically significant aortic regurgitation (AR) who are indicated for TAVR

ELIGIBILITY:
Inclusion Criteria:

1. Subjects >=18 years of age with continuous flow LVAD (cfLVAD) with clinically significant AR1 leading to cfLVAD dysfunction using cfLVAD ASE guidelines that utilize contemporary management strategies for measurement of AR in patients with cfLVAD2,3:

   • AR is graded from 0 to 6 (0 = none; 1 = trace; 2 = mild; 3 = mild-to-moderate; 4 = moderate; 5 = moderate-to-severe; 6 = severe). Considering that AR during continuous flow LVAD (cfLVAD) support is generally both systolic and diastolic, AR is deemed significant if graded ≥ 3.1
2. Patient with NYHA functional class III/IV
3. Patient with high risk for SAVR as documented by Heart Team.
4. Patient has suitable anatomy to accommodate the insertion and delivery of the JenaValve Trilogy™ Heart Valve System
5. Patient or the patient's legal representative has provided written informed consent
6. Patient or the patient's legal representative agrees to comply with all required post-procedure follow-up visits

Exclusion Criteria:

1. Congenital uni- or bicuspid (Sievers 0) aortic valve morphology
2. Previous prosthetic aortic valve (bioprosthesis or mechanical) implant
3. Mitral regurgitation > moderate
4. Clinically significant coronary artery disease (CAD) requiring revascularization within 30 days prior to index procedure, or planned CAD revascularization procedure within 12 months after index procedure
5. Echocardiographic or CT evidence of left ventricular or aortic valve thrombus
6. Ongoing sepsis or active infective endocarditis with ongoing antibiotic (including suppressive) therapy or positive blood cultures within 6 weeks
7. Hypertrophic cardiomyopathy with or without obstruction
8. Severe pulmonary hypertension (systolic PA pressure >80 mmHg)
9. Decompensated right heart failure as assessed clinically and, if available, by baseline right heart catheterization hemodynamics (e.g., right atrial pressure > pulmonary capillary wedge pressure and cardiac index < 2.5 L/min/m2
10. Severe RV dysfunction as assessed clinically and by echocardiography
11. Aortic annular diameter of <21.0 mm or > 28.6 mm (assessed by Multi-detector CT measurement)
12. Aortic annulus angulation > 70° (assessed by Multi-detector CT measurement)
13. Straight length of ascending aorta of < 55 mm
14. Significant disease of ascending aorta, including ascending aortic aneurysm (defined as maximal luminal diameter of 50 mm or greater) or atheroma (including if thick [>5 mm], protruding or ulcerated)
15. Myocardial infarction < 30 days prior to index procedure
16. Cerebrovascular event (TIA, stroke) < 180 days prior to index procedure
17. Blood dyscrasias as defined: leukopenia (WBC < 3000/mm³), or thrombocytopenia (platelets < 90,000/μl) or anemia (Men: Hgb < 8.1 g/dl; Women: Hgb < 7.4 g/dl)
18. Active peptic ulcer or upper gastrointestinal bleeding < 90 days prior to index procedure
19. Known hypersensitivity or contraindication to aspirin, heparin, ticlopidine or clopidogrel, nitinol, tantalum or allergy to contrast agents that cannot be premedicated
20. Subject unable to undergo pre-procedure transesophageal echocardiography or Multi-Detector CT (MDCT) scan for aortic annular sizing
21. Patient is enrolled in another investigational medical device or drug study which has not completed the required primary endpoint follow-up. (Note: Patients involved in a long-term surveillance phase of another study are eligible for enrollment in this registry)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-12-09 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Device Success | 30 days
  Freedom from unsuccessful delivery of the device, and retrieval of the delivery system
Device Positioning | 30 days
  Freedom from incorrect positioning of a single prosthetic heart valve into the proper anatomical location
Device Performance | 30 days
  Intended performance of the valve (i.e., no moderate or severe prosthetic valve regurgitation)*
Surgery/intervention related to device | 30 days
  Freedom from surgery or intervention related to the device# or to a major vascular or access-related or cardiac structural complication
Bleeding | 30 days
  Freedom from VARC type 2-4 bleeding
All Stroke | 30 days
  Number of patients that had stroke
Acute Kidney Injury | 30 days
  Number of patients that had acute kidney injury (AKI) stage 3 or 4
Total aortic regurgitation | 30 days
  Number of patients that had moderate or severe total aortic regurgitation
Major Vascular Complication | 30 days
  Number of patients that had major vascular, access-related, or cardiac structural complication
Permanent pacemaker implantation | 30 days
  Number of patients that had these events
All-cause mortality | 30 days
  All-cause mortality within the first 30 days post index procedure

SECONDARY OUTCOMES:
Device Success | 30 days and 1 year
  Freedom from unsuccessful delivery of the device, and retrieval of the delivery system
Device Positioning | 30 days and 1 year
  Freedom from incorrect positioning of a single prosthetic heart valve into the proper anatomical location
Device Performance | 30 days and 1 year
  Intended performance of the valve (i.e., no moderate or severe prosthetic valve regurgitation)*
Surgery/intervention related to device | 30 days and 1 year
  Freedom from surgery or intervention related to the device# or to a major vascular or access-related or cardiac structural complication
Bleeding | 30 days and 1 year
  Freedom from VARC type 2-4 bleeding
All Stroke | 30 days and 1 year
  Number of patients that had stroke
Acute Kidney Injury | 30 days and 1 year
  Number of patients that had acute kidney injury (AKI) stage 3 or 4
Total aortic regurgitation | 30 days and 1 year
  Number of patients that had moderate or severe total aortic regurgitation
Major Vascular Complication | 30 days and 1 year
  Number of patients that had major vascular, access-related, or cardiac structural complication
Permanent pacemaker implantation | 30 days and 1 year
  Number of patients that had these events
All-cause mortality | 30 days and 1 year
  All-cause mortality within the first 30 days post index procedure

CONTACTS AND LOCATIONS:
Overall Officials: Nir Uriel, MD, Study Chair — Columbia University; Vinod Thourani, MD, Principal Investigator — Piedmont Heart Institute; Ravi Ramana, DO, Principal Investigator — advocate christ medical center; Gabriel Sayer, MD, Principal Investigator — Columbia University
Locations (14):
- United States (14):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - Emory University, Atlanta, Georgia
  - Piedmont, Atlanta, Georgia
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Washington University in St. Louis, St Louis, Missouri
  - Washington University, St. Louis, St Louis, Missouri
  - Columbia University Medical Center/New York-Presbyterian Hospital, New York, New York
  - Houston Methodist Research Center, Houston, Texas
  - Intermountain, Murray, Utah
  - Sentara Norfolk General Hospital, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Uriel N, Sayer G, Addetia K, et al. Hemodynamic Ramp Tests in Patients With Left Ventricular Assist Devices. JACC Heart Fail 2016; 4(3): 208-17. — https://pubmed.ncbi.nlm.nih.gov/26746378/
- See also: Stainback RF, Estep JD, Agler DA, et al. Echocardiography in the Management of Patients with Left Ventricular Assist Devices: Recommendations from the American Society of Echocardiography. J Am Soc Echocardiogr 2015; 28(8): 853-909. — https://pubmed.ncbi.nlm.nih.gov/26239899/
- See also: Accurate Quantification Methods for Aortic Insufficiency Severity in Patients With LVAD: Role of Diastolic Flow Acceleration and Systolic-to-Diastolic Peak Velocity Ratio of Outflow Cannula — https://pubmed.ncbi.nlm.nih.gov/26684975/